CLINICAL TRIAL: NCT07212946
Title: Four Doses of Ayahuasca or Esketamine in Major Depressive Disorder: a Double-blind Randomized Trial
Brief Title: Ayahuasca and Esketamine for Major Depression
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Rafael Guimarães dos Santos, PhD, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 32564020000005440
Record Dates: First submitted 2025-10-01; First posted 2025-10-08 (Actual); Last update posted 2025-12-29 (Actual); Status verified 2025-12

CONDITIONS: Major Depression Severe
MeSH Terms: interventions — Esketamine; Ketamine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ayahuasca (Experimental): oral ayahuasca
  Interventions: Drug: Ayahuasca; Drug: Esketamine
- esketamine (Active Comparator): oral esketamine
  Interventions: Drug: Ayahuasca; Drug: Esketamine

INTERVENTIONS:
Drug: Ayahuasca — Oral
Drug: Esketamine — oral
  Other Names: ketamine

SUMMARY:
Double-blind, randomized trial comparing 4 weekly doses of oral ayahuasca and esketamine in patients with major depression.

ELIGIBILITY:
Inclusion Criteria:

- Clinical diagnosis of depressive disorder

Exclusion Criteria:

- Presence of psychiatric and other medical comorbidities

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2022-10-30 (Actual); Primary Completion 2024-10-30 (Actual); Study Completion 2025-10-01 (Actual)

PRIMARY OUTCOMES:
Beck Depression Inventory | 49 days
  21-question multiple-choice self-report inventory, where higher scores mean worse/more depressive symptoms

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital das Clínicas da FMRP-USP, Ribeirão Preto, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No